CLINICAL TRIAL: NCT00377221
Title: Rectal Health, Behaviors and Microbicide Acceptability
Brief Title: Anorectal Microbicide Project(AMP): Rectal Health, Behaviors and Microbicide Acceptability
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); AIDS Research Alliance (Other); Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Other Study IDs: U19-AI060614:P3 Aim1; 05-07-098; H.34.05.08.24; ARA010; U19AI060614 (NIH)
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Rectal Health; Rectal Behaviors; Anorectal Symptomatology

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Observational, cross-sectional, single-visit study of 896 men and women in Los Angeles, CA and Baltimore, MD including a computer-assisted interview focusing on the behavioral repertoire surrounding RAI, symptoms, and health seeking behaviors and a multidimensional assessment of behaviors, anorectal examination, and testing for sexually transmitted infections (STIs).

ELIGIBILITY:
Inclusion Criteria:

Men and women are eligible who meet all of the following criteria:

1. At least 18 years of age
2. Willing to be tested for STIs including HIV
3. Willing to undergo an anal exam
4. Mentally competent to understand study procedures and give informed consent.
5. For the NO-RAI groups:

   No RAI in the past year for the non-RAI men and women
6. For the practicing RAI groups:

Males: report RAI in the past 30 days Females: report RAI in the past 12 months

Exclusion Criteria:

1. Less than 18 years of age
2. Unwilling to be tested for STIs (and HIV)
3. Unwilling to undergo an anal exam
4. Unwilling to complete study questionnaire
5. Not mentally competent to understand study procedures and give informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 896 (Estimated)
Dates: Start 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: Pamina Gorbach, DrPH, Principal Investigator — University of California, Los Angeles; Peter A Anton, MD, Principal Investigator — University of California, Los Angeles; Ross Cranston, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - AIDS Research Alliance, Los Angeles, California
  - Johns Hopkins University, Baltimore, Maryland